CLINICAL TRIAL: NCT03141398
Title: Continuous Glucose Monitoring (CGM) Versus Oral Glucose Tolerance Test (OGTT) Versus T2* MRI Of The Pancreas In High-Risk Group (Hemoglobinopathies, Lymphoma & Acute Lymphoblastic Leukemia): A Comparative Study
Brief Title: Comparing CGM and OGTT in Relation to Iron Overload Detected by Pancreas T2* MRI in High-Risk Hematology Group
Acronym: CGMs
Status: Withdrawn | Type: Observational
Why Stopped: Due to issues with study design
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16298/16
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-05

CONDITIONS: Iron Overload; Hemoglobinopathies; Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Iron Overload; Hemoglobinopathies; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Continuous Glucose Monitoring; Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- High-Risk Group: The objective of the study to compare the efficiency of detecting glycemic abnormalities using Continuous Glucose Monitoring (CGMs) versus Oral Glucose Tolerance Test (OGTT) and HbA1C. versus T2* MRI of the pancreas (T2* MRI of the Pancreas) in high-risk patients due to insulin deficiency (potential beta cell injury) and those with insulin resistance and to study the different factors that may affect the glycemic control in these patients in relation to their results like the Dose of corticosteroids and chemotherapy in ALL and Hemoglobinopathies,Liver function in ALL and Hemoglobinopathies, and Serum ferritin in Hemoglobinopathies and their transfusion status.
  Interventions: Diagnostic Test: Continuous Glucose Monitoring (CGM); Diagnostic Test: Oral Glucose Tolerance Test (OGTT); Diagnostic Test: T2* MRI of the Pancreas

INTERVENTIONS:
Diagnostic Test: Continuous Glucose Monitoring (CGM) — Where a pager-sized device fixed to the patient's forearm by a diabetic educator and it will connect to his/her body with the sensor, which measures blood glucose for three days. Patients' may experience little pain from needle prick when a sensor is introduced.
Diagnostic Test: Oral Glucose Tolerance Test (OGTT) — Oral glucose tolerance test requires the patient to be fasting and checking of blood sugar after 8 to 10 hours overnight fasting the blood sugar will be checked three times When you arrive to the lab then twice one hour, apart you can have pain due to needle prick or little bleeding at the puncture site.
Diagnostic Test: T2* MRI of the Pancreas — MRI [Magnetic resonance imaging] of the pancreas which is safe and takes around 30 minutes.

SUMMARY:
A prospective, observational, comparative study with no intervention.The objective of the study to compare the efficiency of detecting glycemic abnormalities using Continuous Glucose Monitoring (CGMs) versus Oral Glucose Tolerance Test (OGTT) and HbA1C (Glycated Hemoglobin) and their relation to iron overload detected by T2* MRI of the pancreas in high-risk patients due to insulin deficiency (potential beta cell injury) and those with insulin resistance and to study the different factors that may affect the glycemic control in these patients in relation to their results like the Dose of corticosteroids and chemotherapy in ALL and Hemoglobinopathies, Liver function in ALL and Hemoglobinopathies, and Serum ferritin in Hemoglobinopathies and their transfusion status. Using Validated Tools with Permission, the participants will be selected through probability (random) sampling method with expected subjects numbers ALL/L: 30-50, Thalassemia Major: 20, Sickle cell disease: 20.

ELIGIBILITY:
Inclusion Criteria:

* This study will include participants who are High-risk patients to develop glycemic abnormalities:

  1. Thalassemia major and SCD (beta cell toxicity and hepatic siderosis)
  2. ALL/L ( beta cell injury and hepatic injury due to chemotherapy, and insulin resistance due to corticosteroids)

Exclusion Criteria:

* Age < 14 years;
* Other systemic diseases, renal disorders or malnourished;
* Patients and unwilling to participate in the study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The targeted sample size is up to 100 patients (we aim to recruit approximately 70-100 cases based on the statistics from the outpatient clinics at NCCCR and the cancer registry data; over a period of 3 years). All cases of ALL, Lymphoma, Thalassemia and sickle cell disease diagnosed in HMC will be identified as subjects and they will be recruited based on informed consent and IRB approval.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Efficiency of continuous glucose monitoring compared to oral glucose tolerance and MRI of the Pancreas | 12 Months
  Compare the efficiency of detecting glycemic abnormalities using CGMS versus OGTT vs HbA1C. in high-risk patients due to insulin deficiency (potential beta cell injury) and those with insulin resistance. Detect the prevalence of glycemic abnormalities detected in the same group of patients (high-risk patients) using three different modalities of testing (CGMS, OGTT, HbA1C)and T2*MRI for pancreas

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Yassin, Principal Investigator — Hamad Medical Corporation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gross TM, Bode BW, Einhorn D, Kayne DM, Reed JH, White NH, Mastrototaro JJ. Performance evaluation of the MiniMed continuous glucose monitoring system during patient home use. Diabetes Technol Ther. 2000 Spring;2(1):49-56. doi: 10.1089/152091500316737. PMID 11467320
- [Background] Potts RO, Tamada JA, Tierney MJ. Glucose monitoring by reverse iontophoresis. Diabetes Metab Res Rev. 2002 Jan-Feb;18 Suppl 1:S49-53. doi: 10.1002/dmrr.210. PMID 11921430
- [Background] Bode B, Gross K, Rikalo N, Schwartz S, Wahl T, Page C, Gross T, Mastrototaro J. Alarms based on real-time sensor glucose values alert patients to hypo- and hyperglycemia: the guardian continuous monitoring system. Diabetes Technol Ther. 2004 Apr;6(2):105-13. doi: 10.1089/152091504773731285. PMID 15117576
- [Background] Hoi-Hansen T, Pedersen-Bjergaard U, Thorsteinsson B. Reproducibility and reliability of hypoglycaemic episodes recorded with Continuous Glucose Monitoring System (CGMS) in daily life. Diabet Med. 2005 Jul;22(7):858-62. doi: 10.1111/j.1464-5491.2005.01552.x. PMID 15975099
- [Background] Klonoff DC. Continuous glucose monitoring: roadmap for 21st century diabetes therapy. Diabetes Care. 2005 May;28(5):1231-9. doi: 10.2337/diacare.28.5.1231. No abstract available. PMID 15855600
- [Background] Nichols GA, Hillier TA, Brown JB. Progression from newly acquired impaired fasting glusose to type 2 diabetes. Diabetes Care. 2007 Feb;30(2):228-33. doi: 10.2337/dc06-1392. PMID 17259486
- [Background] Barr EL, Zimmet PZ, Welborn TA, Jolley D, Magliano DJ, Dunstan DW, Cameron AJ, Dwyer T, Taylor HR, Tonkin AM, Wong TY, McNeil J, Shaw JE. Risk of cardiovascular and all-cause mortality in individuals with diabetes mellitus, impaired fasting glucose, and impaired glucose tolerance: the Australian Diabetes, Obesity, and Lifestyle Study (AusDiab). Circulation. 2007 Jul 10;116(2):151-7. doi: 10.1161/CIRCULATIONAHA.106.685628. Epub 2007 Jun 18. PMID 17576864
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2005 Jan;28 Suppl 1:S37-42. doi: 10.2337/diacare.28.suppl_1.s37. No abstract available. PMID 15618111
- [Background] Soliman A, DeSanctis V, Yassin M, Elalaily R, Eldarsy NE. Continuous glucose monitoring system and new era of early diagnosis of diabetes in high risk groups. Indian J Endocrinol Metab. 2014 May;18(3):274-82. doi: 10.4103/2230-8210.131130. PMID 24944918
- [Background] Chen Z, Shen J, Xu LL, Fu XJ, Li JM, Ma YY. [Accuracy of a continuous glucose monitoring system in detection of blood glucose during oral glucose tolerance test]. Nan Fang Yi Ke Da Xue Xue Bao. 2011 Jun;31(7):1256-8. Chinese. PMID 21764709
- [Background] Zhou J, Mo Y, Li H, Ran X, Yang W, Li Q, Peng Y, Li Y, Gao X, Luan X, Wang W, Xie Y, Jia W. Relationship between HbA1c and continuous glucose monitoring in Chinese population: a multicenter study. PLoS One. 2013 Dec 23;8(12):e83827. doi: 10.1371/journal.pone.0083827. eCollection 2013. PMID 24376762
- [Background] He LP, Wang C, Zhong L, Yang YZ, Long Y, Zhang XX, Shu SQ, Yu HL, Yu TT, Wang WP, Wang Y, Ran XW. [Glycemic excursions in people with normal glucose tolerance in Chengdu]. Sichuan Da Xue Xue Bao Yi Xue Ban. 2009 Jul;40(4):704-7. Chinese. PMID 19764578
- [Background] Chen T, Xu F, Su JB, Wang XQ, Chen JF, Wu G, Jin Y, Wang XH. Glycemic variability in relation to oral disposition index in the subjects with different stages of glucose tolerance. Diabetol Metab Syndr. 2013 Jul 23;5:38. doi: 10.1186/1758-5996-5-38. eCollection 2013. PMID 23876034